CLINICAL TRIAL: NCT05069051
Title: BeliVeR a Phase II Trial of Belimumab in Combination with Rituximab/venetoclax in Patients with Refractory or Relapsed Chronic Lymphocytic Leukemia
Brief Title: Belimumab in Patients with Chronic Lymphocytic Leukemia
Acronym: BeliVeR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeliVeR, 3.0, 12.11.2021
Record Dates: First submitted 2021-09-09; First posted 2021-10-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Chronic Lymphoid Leukemia in Relapse
Keywords: relapsed CLL; refractory CLL
MeSH Terms: interventions — belimumab; Standard of Care

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, two-armed controlled, multicenter phase II study analyzing the efficacy and safety of belimumab in combination with venetoclax plus rituximab in patients with refractory or relapsed CLL.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Belimumab (Experimental): Patients obtain belimumab in combination with rituximab/venetoclax
  Interventions: Drug: Belimumab 200 MG/ML [Benlysta]
- Standard of Care (Active Comparator): Patients obtain the combination rituximab/venetoclax
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: Belimumab 200 MG/ML [Benlysta] — Patients obtain belimumab treatment in combination with rituximab and venetoclax
  Arms: Belimumab
Drug: standard of care — Patients obtain the standard of care: combination rituximab and venetoclax
  Arms: Standard of Care

SUMMARY:
This study is a phase II trial of belimumab in combination with rituximab/venetoclax in patients with refractory or relapsed chronic lymphocytic leukemia (CLL). Treatment of CLL has drastically changed in the past years as new therapeutic agents have gained clinical approval. The combination rituximab/venetoclax over a course of two years is approved as second line therapy especially in patients with high risk CLL (del17p), showing high remission rates and achievement of MRD (minimal residual disease) negativity. The next goals in CLL therapy are now to increase the rate of MRD negativity and to achieve an earlier MRD negativity during the course of treatment to allow for a reduction of treatment time and therefore treatment-induced toxicities. In line with other hematologic diseases, progression free survival depends on remission status, especially MRD negativity, after last treatment as MRD positivity after therapy indicates the persistence of treatment resistant CLL cells. One mechanism of therapy resistance has been described as reduced sensitivity to rituximab-induced antibody dependent cell-mediated cytotoxicity (ADCC) by natural killer (NK) cell production of B-lymphocyte stimulator (BlyS, also called BAFF), which can be bound by belimumab, a human anti-BAFF antibody. Moreover, recombinant human (rh)BAFF can dose dependently reverse cytotoxic effects of venetoclax, which could also be restored by the application of belimumab. This led to the conceptualization of this clinical trial, in which belimumab is applied as a weekly subcutaneous injection in combination with standardrituximab/venetoclax treatment for up to 24 months in relapsed and refractory CLL patients. By removing BAFF from the CLL microenvironment we aim to increase the efficacy of rituximab/venetoclax treatment to achieve higher and earlier MRD negativity rates and allow for an abbreviated treatment.

DETAILED DESCRIPTION:
The treatment landscape for relapsed/refractory CLL has faced profound changes and new developments in the past years. Conventional chemoimmunotherapies show only limited efficacy in the relapsed setting and are associated with side effects caused by rather unspecific mode of action of chemotherapy. Therefore, several targeted agents have become available for the treatment of CLL in recent years. However, beside the combination of rituximab and venetoclax all of these substances require continuous treatment bearing the risk of developing therapy resistance and accumulation of side effects. The combination of rituximab and venetoclax shows high response rates in the relapsed setting with MRD negativity rates of 83%, however still requiring a 2-year period of continuous treatment. Future efforts have now to focus on the further and earlier elimination of MRD in all treated patients to allow for a reduced treatment time and therefore lower risks of side effects and development of resistance as well as the achievement of long-lasting remission and potential cure in the future. The available data on the sensitizing effect of belimumab for venetoclax treatment, together with the published results showing a belimumab-induced sensitization of CLL cells to NK cell antitumor immunity as mediated by rituximab, provide a clear rationale for the evaluation of a combinatorial treatment with belimumab to increase sensitivity and response to the established CLL treatment regimen venetoclax/rituximab. Thus, we here propose an open-label, randomized, controlled, multicenter Phase II study analyzing safety and efficacy of belimumab in combination with venetoclax and rituximab in patients with refractory or relapsed CLL.

Justification of combinational treatment The published and preclinical data on the sensitizing effect of belimumab on CLL cells to venetoclax and rituximab provides a clear rationale for combinational treatment of rituximab/venetoclax with belimumab. Although high MRD negativity rates are achieved withrituximab/venetoclax some patients still present with persisting MRD and suffer from early disease relapse. This phase II trial is designed to investigate the efficacy of belimumab in addition to rituximab/venetoclax in relapsed/refractory CLL. The primary endpoint is achievement of MRD negativity at end of induction treatment (EOI). Furthermore, the following secondary objectives will be assessed:

* Safety of belimumab and rituximab/venetoclax in patients with relapsed or refractory CLL
* Overall response rate (ORR)
* Progression free survival (PFS)
* Overall survival (OS)
* Duration of response (DOR)
* Assessment of further efficacy markers of belimumab in combination with rituximab/venetoclax in CLL compared to control
* Pharmacokinetics of belimumab in CLL patients

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* Diagnosis of CLL/SLL established according to iwCLL criteria
* Refractory or relapsed CLL that warrants treatment (according to modified criteria for initiation of therapy (Hallek et al., 2018)):

  1. Massive (ie, lower edge of spleen ≥6 cm below the left costal margin), progressive, or symptomatic splenomegaly, or
  2. Massive (ie, ≥10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy, or
  3. Progressive lymphocytosis in the absence of infection, with an increase in blood ALC≥50% over a 2-month period or lymphocyte doubling time of <6 months (as long as initial ALC was ≥30,000/L), or
  4. Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy, or
  5. Constitutional symptoms, defined as any one or more of the following disease-related symptoms or signs occurring in the absence of evidence of infection:

     * Unintentional weight loss of ≥10% within the previous 6 months, or
     * Significant fatigue (≥Grade 2), or
     * Fevers >38.0°C for ≥2 weeks, or
     * Night sweats for >1 month.
* CLL relapsing after any line of treatment that included radiotherapy, chemotherapy, immunotherapy, or small molecules. Patients who relapse after a previous therapy with venetoclax can be included in the study in case of a late relapse (i.e. >18 months after venetoclax was discontinued.
* Discontinuation of all therapy (including radiotherapy, chemotherapy, immunotherapy, or small molecules) for the treatment of CLL ≥2 weeks before study treatment excluding systemic corticosteroids for symptomatic control.
* All acute toxic effects of any prior antitumor therapy resolved to Grade ≤1 before treatment (with the exception of alopecia [Grade 1 or 2 permitted], neurotoxicity [Grade 1 or 2 permitted], or bone marrow parameters [any of Grade 1, 2, 3, or 4 permitted).
* Eastern Cooperative Oncology Group [ECOG] < 3.
* Required baseline laboratory data (within 4 weeks prior to treatment):
* Serum total bilirubin ≤1.5 x ULN (unless directly attributable to CLL disease or to Gilbert's Syndrome)
* ALT/AST ≤2.5 x ULN
* Renal creatinine clearance >30 ml/min
* Neutrophile count >1.000/μl (unless directly attributable to CLL disease)
* Negative serological Hepatitis B and C test or negative PCR in case of positive serological test without evidence of an active infection, negative HIV test within 6 weeks prior to treatment.
* Written informed consent of the subject after clarification

Exclusion Criteria:

* (Suspicion of) transformation of CLL (i.e. Richter's transformation, pro-lymphocytic leukemia) or central nervous system (CNS) involvement
* IgG < 4 g/L under substitution of immunoglobulins
* Early relapse (i.e <18 months) after any line of treatment that included venetoclax.
* Malignancies other than CLL currently requiring systemic therapies
* Evidence of active systemic bacterial (e.g. tuberculosis), fungal, or viral infection (e.g., CMV) at the time of initiation of therapy
* Confirmed progressive multifocal leukencephalopathy (PML)
* Known history of drug-induced liver injury (DILI), chronic/active hepatitis C (HCV), chronic/active hepatitis B (HBV)
* Requirement of therapy with strong CYP3A4 inhibitors/ inducers or anticoagulant with phenprocoumon or other vitamin K-antagonists
* Active inflammatory bowel disease
* History of prior allogeneic bone marrow or organ transplantation
* Ongoing immunosuppressive therapy. Subjects may use topical, enteric, or inhaled corticosteroids as therapy for comorbidities and systemic steroids for autoimmune anemia and/or thrombocytopenia. Ongoing use of low-dose systemic corticosteroids (≤5 mg/day of methylprednisolone or equivalent) for rheumatologic conditions is permitted
* History of primary immunodeficiency
* Concurrent participation in another therapeutic clinical trial
* History of serious suicide risk including any suicidal behaviour in the last 6 months
* Live vaccination 30 days prior to treatment
* Hypersensitivity known from medical history to one of the drugs used or their ingredients or to drugs with a similar chemical structure
* Simultaneous participation in another interventional clinical trial (including within the last 4 weeks before inclusion)
* Addictions or other illnesses that do not allow the person concerned to assess the nature and extent of the clinical trial and its possible consequences
* Pregnant or breastfeeding women
* Women of childbearing potential, except women who meet the following criteria:

  * post-menopausal (12 months natural amenorrhoea or 6 months amenorrhoea with serum FSH > 40 U/ml)
  * postoperative (6 weeks after bilateral ovarectomy with or without hysterectomy)
  * regular and correct use of a contraceptive method with an Pearl Index < 1% per year, which will have to be continued for up to four months after the discontinuation of the study drug
  * sexual abstinence
  * Vasectomy of the partner
* Male subjects who are able to father a child, except men who meet the following criteria:

  * willingness to abstain from heterosexual intercourse or use a protocolrecommended method contraception from the screening visit throughout the study treatment period and for 90 days following the last dose of study drug
  * refrain from sperm donation from screening visit throughout the study treatment period and for four months following the last dose of study drug
* Indications that the subject is unlikely to adhere to the protocol (e.g., lack of compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-07-14 (Estimated)

PRIMARY OUTCOMES:
Negativity rate of minimal residual disease (MRD) in peripheral blood (PB) measured by flow cytometry at EOI | Baseline, Day 1
  MRD negativity is defined as less than one CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. The MRD negativity rate is defined as the proportion of patients having achieved MRD negativity. Patients without any evaluable MRD sample at end of induction treatment will be kept and labeled as 'MRD positive (≥10-4)' in the analysis.
Negativity rate of minimal residual disease (MRD) in peripheral blood (PB) measured by flow cytometry at EOI | During the intervention: Cycle 1 Day 1, (Cycle length 15 days)
  MRD negativity is defined as less than one CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. The MRD negativity rate is defined as the proportion of patients having achieved MRD negativity. Patients without any evaluable MRD sample at end of induction treatment will be kept and labeled as 'MRD positive (≥10-4)' in the analysis.
Negativity rate of minimal residual disease (MRD) in peripheral blood (PB) measured by flow cytometry at EOI | During the intervention: Cycle 4 Day 1 (Cycle length 15 days)
  MRD negativity is defined as less than one CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. The MRD negativity rate is defined as the proportion of patients having achieved MRD negativity. Patients without any evaluable MRD sample at end of induction treatment will be kept and labeled as 'MRD positive (≥10-4)' in the analysis.
Negativity rate of minimal residual disease (MRD) in peripheral blood (PB) measured by flow cytometry at EOI | During 4 weeks after Cycle 6 Day 1 (Cycle length 15 days)
  MRD negativity is defined as less than one CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. The MRD negativity rate is defined as the proportion of patients having achieved MRD negativity. Patients without any evaluable MRD sample at end of induction treatment will be kept and labeled as 'MRD positive (≥10-4)' in the analysis.
Negativity rate of minimal residual disease (MRD) in peripheral blood (PB) measured by flow cytometry at EOI | End of treatment: 2 years after Cycle 1 at Day 2 (Cycle length 15 days)
  MRD negativity is defined as less than one CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. The MRD negativity rate is defined as the proportion of patients having achieved MRD negativity. Patients without any evaluable MRD sample at end of induction treatment will be kept and labeled as 'MRD positive (≥10-4)' in the analysis.
Negativity rate of minimal residual disease (MRD) in peripheral blood (PB) measured by flow cytometry at EOI | Follow-Up: every 3 months up to 1 year
  MRD negativity is defined as less than one CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. The MRD negativity rate is defined as the proportion of patients having achieved MRD negativity. Patients without any evaluable MRD sample at end of induction treatment will be kept and labeled as 'MRD positive (≥10-4)' in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Walz, Prof.Dr., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, CCU Translational Immunology, Tübingen, Baden-Wurttemberg, Germany